CLINICAL TRIAL: NCT04902313
Title: Cultivating Resilience in Oncology Practice: A Feasibility Study of Pediatric Patients
Brief Title: Cultivating Resilience in Oncology Practice
Acronym: CROP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Oskar Lundgren, MD, PhD, MSc, Lecturer, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-01044
Record Dates: First submitted 2021-04-23; First posted 2021-05-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2021-05

CONDITIONS: Childhood Cancer; Depressive Symptoms; Anxiety Disorders and Symptoms; Mental Health Issue
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Interventional group of cancer patients, and observational group of pediatric patients with other chronic conditions.
Who Masked: Outcomes Assessor
Masking Description: Collection of data and analysis will be made by researcher with limited knowledge of participant status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer patients (Experimental): Youths (10-18 y) with newly diagnosed cancer, as well as their family members.
  Interventions: Behavioral: Awareness and insight Modules (AiM)
- Pediatric patients (Active Comparator): Youths (10-18 y) with a chronic somatic disease receiving care at a pediatric outpatient facility.
  Interventions: Behavioral: Awareness and insight Modules (AiM)

INTERVENTIONS:
Behavioral: Awareness and insight Modules (AiM) — 12 week of daily reflection and meditation exercises, delivered by mobile phone text messages, after 3-4 live introduction sessions.

SUMMARY:
The purpose of the CROP study is to investigate the potential to cultivate psychological resources and resilience in childhood cancer patients and their family members using a mobile phone-based intervention.

The feasibility study aims to evaluate the implementation and participant experience of the digital intervention and register psychological outcome measures preliminary evidence for its acceptability, feasibility, and potential beneficial effects.

DETAILED DESCRIPTION:
The feasibility study (CROP) will recruit 20 youths with newly diagnosed cancer (10-18 y) and family members for participation in a 12-week digital intervention to cultivate psychological resources.

Investigators will recruit an equal number of pediatric patients with other chronic conditions to an observational comparison group to indicate the influences on participation and outcome from the oncology care context.

Investigators will obtain informed consent from all participants. Upon inclusion in the study, participants will start getting a text message every day for 12 consecutive weeks. The texts will contain links to a digital platform on which participants will complete an exercise in either self-reflection or guided mindfulness meditation.

The psychological training program is based on 12 modules with evidence-based treatments in other medical contexts and age groups. The practices are based on acceptance, commitment, re-appraisal, meaning and purpose, expressive writing, narrative processes, mindfulness, compassion, equanimity, and gratitude. The combination of practices and the implementation in pediatric oncology has not been studied earlier.

The cancer patients will be recruited during the first month after diagnosis, meet with an instructor during 2-4 start-up meetings, and thereafter practice on their own or with participating family members.

The pediatric patients with chronic diseases will be recruited during a follow-up visit to an out-patient clinic and meet with an instructor during 2-4 start-up meetings, and thereafter practice on their own or together with participating family members.

Investigators will address the primary research question of the feasibility of the intervention by investigating participant activity data, written evaluations of the experience of participation, and through phone interviews of participants.

Secondary research questions, such as preliminary data on changes in mental health and psychological distress, will be investigated with self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cancer
* Chronic pediatric disease

Exclusion Criteria:

* Severe crisis reaction
* Late-stage palliative care
* Severe intellectual disability
* Psychiatric disease hindrance
* Participation in other study with psychological intervention

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Mental Health Continuum-Short Form (MHC-SF) | At the beginning of the trial.
  14 items. Score (min-max): 0-70. A high score indicates mental well-being.
Mental Health Continuum-Short Form (MHC-SF) | After 12 weeks of participation in the trial.
  14 items. Score (min-max): 0-70. A high score indicates mental well-being.
Mental Health Continuum-Short Form (MHC-SF) | At 12-month after completion of the trial.
  14 items. Score (min-max): 0-70. A high score indicates mental well-being.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) | At the beginning of the trial.
  25 items. Score (min-max): 0-25. A high score indicates psychiatric difficulties.
Strenghs and Difficulties Questionnaire (SDQ) | After 12 weeks of participation in the trial.
  25 items. Score (min-max): 0-25. A high score indicates psychiatric difficulties.
Strengths and Difficulties Questionnaire (SDQ) | At 12-month after completion of the trial.
  25 items. Score (min-max): 0-25. A high score indicate psychiatric difficulties.
Revised Child Anxiety and Depression Scale Short form (RCADS-SF) | At the beginning of the trial.
  25 items. Score (min-max): 0-75. A high score indicates symptoms of anxiety and depression.
Revised Child Anxiety and Depression Scale (RCADS) | After 12 weeks of participation in the trial.
  25 items. Score (min-max): 0-75. A high score indicates symptoms of anxiety and depression.
Revised Child Anxiety and Depression Scale (RCADS) | At 12-month after completion of the trial.
  25 items. Score (min-max): 0-75. A high score indicates symptoms of anxiety and depression.
System Usability Scale (SUS) | After completion of the 12 week trial.
  10 items. Score (min-max): 10-50. A high score indicates a high level of usability.

CONTACTS AND LOCATIONS:
Overall Officials: Catrin Furuhjelm, MD, PhD, Study Chair — Region Östergötland
Locations (1):
- H.K.H. Crown Princess Victoria Children's Hospital, Linköping University Hospital, Sweden, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Study data will be made available upon reasonable request from other researchers.